CLINICAL TRIAL: NCT05809011
Title: A Multicenter, Randomized, Open-label, Controlled Study to Evaluate the Efficacy and Safety of corticoSTEROids Added to Standard Therapy in Patients With Acute Heart Failure (STERO-AHF)
Brief Title: Efficacy and Safety of corticoSTEROids Added to Standard Therapy in Patients With Acute Heart Failure (STERO-AHF)
Acronym: STERO-AHF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Matteo Pagnesi, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP5676; 2022-003206-69 (EudraCT Number)
Record Dates: First submitted 2023-03-19; First posted 2023-04-12 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; Diuretic resistance; Inflammation; Corticosteroids; Diuretic response
MeSH Terms: conditions — Inflammation | interventions — Dexamethasone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticosteroid therapy plus standard-of-care (Experimental): Patients randomized to this arm will receive a single-bolus intravenous injection of dexamethasone 20 mg at day 1 (as soon as possible after randomization), followed by oral prednisone 1 mg/kg daily (maximum 60 mg daily) from day 2 to day 7 after randomization. Patients randomized to this arm will also receive standard-of-care therapy for acute heart failure.
  Interventions: Drug: Dexamethasone; Drug: Prednisone
- Standard-of-care (No Intervention): Patients randomized to this arm will receive standard-of-care therapy for acute heart failure.

INTERVENTIONS:
Drug: Dexamethasone — After enrollment and randomization, the intervention (experimental arm) will be the administration of corticosteroid therapy, added to standard therapy for acute heart failure. Corticosteroid therapy will be administered as a single-bolus intravenous injection of dexamethasone 20 mg (day 1, as soon as possible after randomization), followed by oral prednisone 1 mg/kg daily (maximum 60 mg daily) from day 2 to day 7 after randomization, administered at about 8.00 AM.
  Arms: Corticosteroid therapy plus standard-of-care
Drug: Prednisone — After enrollment and randomization, the intervention (experimental arm) will be the administration of corticosteroid therapy, added to standard therapy for acute heart failure. Corticosteroid therapy will be administered as a single-bolus intravenous injection of dexamethasone 20 mg (day 1, as soon as possible after randomization), followed by oral prednisone 1 mg/kg daily (maximum 60 mg daily) from day 2 to day 7 after randomization, administered at about 8.00 AM.
  Arms: Corticosteroid therapy plus standard-of-care

SUMMARY:
STERO-AHF is a pilot, prospective, multicenter, randomized, open-label, controlled study aimed to evaluate the diuretic efficacy and early clinical benefit of corticosteroid therapy administered for 7 days, in addition to standard therapy, in patients hospitalized for acute heart failure (AHF) and with evidence of insufficient diuretic response. Eligible patients will be randomized 1:1 to receive either standard-of-care alone (control group) or standard-of-care plus corticosteroid therapy (experimental group) for up to 7 days. Patients will be followed to 30 days.

DETAILED DESCRIPTION:
STERO-AHF is a pilot, prospective, multicenter, randomized, open-label, controlled clinical trial designed to evaluate the efficacy, safety and tolerability of corticosteroid therapy administered for 7 days, when added to standard therapy, in patients with acute heart failure (AHF) and evidence of insufficient diuretic response. After assessing eligibility for the study (screening period), eligible patients will be randomized 1:1 to receive either standard-of-care alone (control group) or standard-of-care plus corticosteroid therapy (experimental group) for up to 7 days.

Study candidates will be adult patients who fulfill the following key inclusion criteria: 1) hospitalized with a primary diagnosis of AHF, either de novo or decompensated chronic heart failure (HF), regardless of left ventricular ejection fraction; 2) insufficient diuretic response at 2-6 hours after the first intravenous loop diuretic dose administration; 3) persistent dyspnea at rest or after mild exertion and clinical signs of fluid overload; 4) elevated C-reactive protein ≥ 10 mg/L at hospital admission. Patients with systolic blood pressure <90 mmHg at time of screening and with severe renal impairment defined as estimated glomerular filtration rate <20 mL/min/1.73m2 or need of chronic dialysis or temporary renal replacement therapy will be excluded from the study.

After enrollment and randomization, patients assigned to corticosteroid therapy will receive it as a single-bolus intravenous injection of dexamethasone 20 mg (day 1), followed by oral prednisone 1 mg/kg daily (maximum 60 mg daily) from day 2 to day 7 after randomization. All enrolled subjects will receive standard-of-care therapy for AHF, including tailored diuretic therapy according to current management strategies for patients with insufficient diuretic response after intravenous loop diuretic dose administration.

The study aim is to evaluate the diuretic efficacy and early clinical benefit of corticosteroid therapy administered for 7 days, when added to standard therapy, in diuretic-resistant patients with AHF. All randomized patients will be assessed daily while hospitalized up to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8), and then will be followed-up at a scheduled visit at 30 days.

The primary endpoints will be assessed at day 8 after randomization or at discharge (in patients discharged earlier than day 8) or at the occurrence of death (in patients dying before day 8). For the safety evaluation, all adverse events will be collected from signing of the informed consent form through day 30. The duration of enrollment will be of ~24 months. The primary completion of the study is the date when the last enrolled patient is assessed for the collection of the primary endpoint. The end of the study is the date when the last enrolled patient has completed the last follow-up visit.

A total of 9 Italian high-volume, tertiary-care centers will be involved in the study. Based on sample size calculations, the trial is targeted to enroll 120 patients with AHF to provide sufficient statistical power to detect a significant difference in diuretic response (primary endpoint).

ELIGIBILITY:
Inclusion criteria:

1. Full age of consent at screening (at least ≥18 years old according to local legislation).
2. Able to provide written informed consent or a legally authorized representative is able to provide written informed consent.
3. Hospitalized for AHF, either de novo or decompensated chronic HF, regardless of LVEF.
4. Treatment with a minimum single dose of 40 mg of intravenous furosemide or equivalent intravenous loop diuretic dose (defined as 20 mg of torsemide or 1 mg of bumetanide) at any time between presentation and the end of screening.
5. Insufficient diuretic response assessed at 2-6 hours after the first intravenous loop diuretic dose administration, according to the latest 2021 ESC guidelines on the management of acute and chronic HF, defined as either urinary sodium <70 mEq/L at a single spot urinary sodium analysis performed at 2 hours or an average urine output <150 mL/h in the first 6 hours after first intravenous diuretic administration. In case of early insufficient diuretic response and persistence of congestion, the dose of intravenous loop diuretic will have to be doubled and the patient may be enrolled.
6. New York Heart Association functional class II, III or IV at screening.
7. Elevated NT-proBNP ≥1400 pg/mL or BNP ≥350 pg/mL according to the local laboratory for patients without atrial fibrillation, or NT-proBNP ≥2200 pg/mL or BNP ≥550 pg/mL for patients with atrial fibrillation at the time of admission and/or in the 72 hours prior to hospital admission.
8. Elevated CRP ≥10 mg/L according to the local laboratory, measured during the current hospitalization.
9. Eligible for randomization within the first 24 hours from presentation.

Exclusion criteria:

1. Dyspnea due to non-cardiac causes.
2. Systolic blood pressure <90 mmHg or >180 mmHg at time of screening and randomization.
3. Current hospitalization for AHF primarily caused by pulmonary embolism, cerebrovascular event, or acute myocardial infarction.
4. Current hospitalization for AHF not caused primarily by volume overload; for example, triggered by significant arrhythmia (e.g., sustained ventricular tachycardia [VT], or atrial fibrillation/flutter with sustained ventricular response >120 beats per minute, or bradycardia with sustained ventricular rate <45 beats per minute), infection/sepsis, severe anemia, uncorrected thyroid disease, or acute exacerbation of chronic obstructive pulmonary disease.
5. Temperature >38.0 °C (oral or equivalent), sepsis, septic shock, or evidence of active infection (either bacterial, fungal or viral) requiring new oral or intravenous anti-microbial treatment (either antibacterial, antifungal or antiviral therapy).
6. History of chronic infections, latent infections, chronic inflammatory or immunosuppressive disorders, chronic immunosuppressive therapy, ongoing chemotherapy or immunotherapy, or chronic anti-microbial therapy (either prophylactic or suppressive).
7. Current treatment with intravenous corticosteroids or chronic oral corticosteroid therapy for any other condition and of any duration in the past 6 months prior to randomization.
8. Documented active or history of hypocortisolism or hypercortisolism caused by primary/secondary adrenal gland disorders, pituitary disorders, iatrogenic conditions, or genetic forms (e.g., adrenal insufficiency, Cushing disease or Cushing syndrome, prior chronic long-standing corticosteroid therapy).
9. Decompensated diabetes mellitus, defined as the presence of diabetic ketoacidosis, hyperglycemic hyperosmolar state, or glycemia > 250 mg/dL as measured at the latest local laboratory exams performed during hospitalization.
10. Acute coronary syndrome / myocardial infarction, stroke, transient ischemic attack, or intracranial bleeding in the past 90 days prior to randomization.
11. Any of the following major interventions performed in the past 30 days prior to randomization or planned during the current admission: major cardiac surgery (e.g., coronary artery bypass graft or valve replacement), percutaneous coronary intervention, transcatheter aortic valve replacement, or percutaneous mitral valve repair (e.g., transcatheter edge-to-edge mitral valve repair); implantation of a cardiac resynchronization therapy device; implantation of a mechanical circulatory support (MCS) device; carotid artery disease revascularization (percutaneous intervention or surgery); or any other surgical procedure that is considered "major" according to investigator judgement.
12. Heart transplant recipient, or listed for heart transplant with expectation to receive transplant during the study period (according to investigator judgement), or currently using or planned for implantation of left ventricular assist device or intra-aortic balloon pump or any other MCS device, or planned inotropic support in an outpatient setting, or planned for palliative care for HF.
13. Hemodynamically significant (severe) uncorrected primary cardiac valvular disease planned for intervention during the study period. Secondary mitral regurgitation or tricuspid regurgitation due to dilated cardiomyopathy is not excluded unless planned for surgical or percutaneous intervention during the study period.
14. AHF caused by peripartum cardiomyopathy or Tako-tsubo syndrome diagnosed within the past 6 months, active myocarditis, or other acute structural heart disease (e.g., acute mitral cord rupture).
15. Cardiomyopathy due to infiltrative diseases (e.g., amyloidosis), accumulation diseases (e.g., haemochromatosis, Fabry disease), hypertrophic obstructive cardiomyopathy, complex congenital heart diseases, or known pericardial constriction.
16. Invasive mechanical ventilation at time of screening (endotracheal intubation). Continuous or intermittent non-invasive mechanical ventilation is allowed.
17. Symptomatic VT in patients without an implantable cardioverter defibrillator in the past 90 days prior to randomization.
18. Symptomatic bradycardia with a documented heart rate <50 beats per minute at electrocardiogram performed before randomization or evidence of advanced atrio-ventricular block (third-degree or second-degree type 2) without a pacemaker.
19. Atrial fibrillation/flutter with a documented, persistent resting heart rate >120 beats per minute at electrocardiogram performed before randomization.
20. Severe impairment of renal function, defined as eGFR <20 mL/min/1.73m2 (according to the CKD-EPI equation) as measured at the latest local laboratory exams performed during hospitalization (between presentation and the end of screening), or requiring chronic dialysis or temporary renal replacement therapy.
21. Acute contrast-induced nephropathy.
22. Severe anemia, defined as hemoglobin <8 g/dL as measured at the latest local laboratory exams performed during hospitalization.
23. Any major solid organ transplant recipient or planned organ transplant during the study period.
24. Known history of glaucoma.
25. Prior gastrointestinal surgery or gastrointestinal disorder that could interfere with the absorption of the study drug (according to investigator judgement).
26. Documented active or suspected malignancy or history of malignancy of any organ system within 1 year prior to screening, except appropriately treated localized basal cell carcinoma of the skin.
27. Presence of any disease other than HF with life expectancy less than 6 months.
28. Decision for palliative care in HF (informed patient decision to adhere to limited HF treatments only).
29. Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial, or less than five half-lives of the study drug (whichever is longer) in case of drug trial. Patients participating in a purely observational study will not be excluded.
30. Known allergy or hypersensitivity to any corticosteroid or any excipient of the study drug product.
31. Chronic alcohol or drug abuse or any condition that makes the patient unreliable or unlikely to complete the trial (according to investigator judgement).
32. Inability to follow instructions or comply with follow-up procedures.
33. Pregnant or nursing (lactating) women. Women of child-bearing potential must have a negative urine or serum pregnancy test prior to enrollment.
34. Any other medical condition that may put the patient at risk or influence study results according to the investigator judgement, or that the investigator deems unsuitable for the study.
35. Inability to comply with all study requirements, due to major comorbidities that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diuretic response, defined as absolute body weight change per 40 mg total dose of intravenous furosemide or equivalent | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  Absolute change in body weight (in kg) per 40 mg total dose of intravenous furosemide or equivalent over the preceding days of the study (equivalent intravenous doses: bumetanide 1 mg, torsemide 20 mg).
Early clinical benefit, defined as a hierarchical composite outcome including all-cause death, worsening heart failure (HF), and the absolute change in patient-reported dyspnea as quantified by the visual analogue scale (VAS) score (0-100 mm scale) | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  All-cause death is defined as the occurrence of death from any cause.
  Worsening HF is defined as worsening signs and/or symptoms of HF that require an intensification of intravenous therapy for HF or mechanical ventilatory, renal or circulatory support. Such treatment can include the introduction or up-titration of intravenous diuretics, intravenous nitrates, intravenous inotropes, intravenous vasoactive agents or any other intravenous therapy for HF, or institution of mechanical support such as mechanical ventilation, ultrafiltration, hemodialysis, intra-aortic balloon pumping or ventricular assist device, etc.
  The absolute change in patient-reported dyspnea is quantified according to the VAS scoring system, a 0-100 mm scale that rates the absolute degree of dyspnea. Patients rate their level of dyspnea on a linguistically-validated scale that rates from 0 to 100, with 0 representing the worst conceivable dyspnea and 100 representing the best imaginable ability to breathe.

SECONDARY OUTCOMES:
Hierarchical composite outcome of all-cause death, total number of heart failure (HF) events, and absolute change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (KCCQ-TSS) | At day 30
  HF event is defined as a hospitalization, an Emergency Department visit, an urgent care visit or an outpatient visit with all the following criteria met: hospitalization or visit due to a primary diagnosis of HF or worsening of HF; at least one symptom of HF; at least two physical examination findings of HF or at least one physical examination finding plus one positive diagnostic test of HF; intensification of therapy for HF.
  KCCQ-TSS is a well-established tool to evaluate health status and quality-of-life in patients with HF. KCCQ is a 23-item, self-administered health status measure for the quantification of HF-related health status. The domains quantified by the KCCQ include physical limitation, symptoms, self-efficacy, quality-of-life, and social limitation. The TSS quantifies symptom frequency and severity and ranges from 0 to 100, with higher score indicating better function.
Absolute change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (KCCQ-TSS) | From baseline to day 30
  KCCQ-TSS is a well-established tool to evaluate health status and quality-of-life in patients with HF. KCCQ is a 23-item, self-administered health status measure for the quantification of HF-related health status. The domains quantified by the KCCQ include physical limitation, symptoms, self-efficacy, quality-of-life, and social limitation. The TSS quantifies symptom frequency and severity and ranges from 0 to 100, with higher score indicating better function.
Improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (KCCQ-TSS) of ≥5 points | At day 30
  KCCQ-TSS is a well-established tool to evaluate health status and quality-of-life in patients with HF. KCCQ is a 23-item, self-administered health status measure for the quantification of HF-related health status. The domains quantified by the KCCQ include physical limitation, symptoms, self-efficacy, quality-of-life, and social limitation. The TSS quantifies symptom frequency and severity and ranges from 0 to 100, with higher score indicating better function.
Absolute change in log-transformed N-terminal pro-B-type natriuretic peptide (NT-proBNP) level | From baseline to day 30
  NT-proBNP is measured in pg/mL
Daily urinary output per daily loop diuretic dose | At day 4 or at the occurrence of death (in patients dying before day 4)
  Daily urine output is measured in mL or L.
  Daily loop diuretic dose is defined as the daily dose (in mg) of oral or intravenous loop diuretics converted to furosemide equivalents: 1 mg bumetanide = 20 mg torsemide = 80 mg furosemide for oral diuretics; 1 mg bumetanide = 20 mg torsemide = 40 mg furosemide for intravenous diuretics. The oral loop diuretic dose is considered to be half the intravenous loop diuretic dose.
Daily urinary output per daily loop diuretic dose | At day 8 or at discharge (in patients discharged earlier than day 8) or at the occurrence of death (in patients dying before day 8)
  Daily urine output is measured in mL or L.
  Daily loop diuretic dose is defined as the daily dose (in mg) of oral or intravenous loop diuretics converted to furosemide equivalents: 1 mg bumetanide = 20 mg torsemide = 80 mg furosemide for oral diuretics; 1 mg bumetanide = 20 mg torsemide = 40 mg furosemide for intravenous diuretics. The oral loop diuretic dose is considered to be half the intravenous loop diuretic dose.
Absolute change in serum creatinine | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  Serum creatinine is measured in mg/dL
Absolute change in estimated glomerular filtration rate (eGFR), calculated according to the CKD-EPI equation | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  eGFR is measured in mL/min/1.73 m2

OTHER OUTCOMES:
Change in patient-reported dyspnea as quantified by the area under the curve (AUC) of daily visual analogue scale (VAS) scores (0-100 mm scale) | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  The absolute change in patient-reported dyspnea is quantified according to the VAS scoring system, a 0-100 mm scale that rates the absolute degree of dyspnea. Patients rate their level of dyspnea on a linguistically-validated scale that rates from 0 to 100, with 0 representing the worst conceivable dyspnea and 100 representing the best imaginable ability to breathe.
Absolute change in patient-reported dyspnea visual analogue scale (VAS) score | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
  The absolute change in patient-reported dyspnea is quantified according to the VAS scoring system, a 0-100 mm scale that rates the absolute degree of dyspnea. Patients rate their level of dyspnea on a linguistically-validated scale that rates from 0 to 100, with 0 representing the worst conceivable dyspnea and 100 representing the best imaginable ability to breathe.
Worsening heart failure (HF) | At day 8
  Worsening HF is defined as worsening signs and/or symptoms of HF that require an intensification of intravenous therapy for HF or mechanical ventilatory, renal or circulatory support. Such treatment can include the introduction or up-titration of intravenous diuretics, intravenous nitrates, intravenous inotropes, intravenous vasoactive agents or any other intravenous therapy for HF, or institution of mechanical support such as mechanical ventilation, ultrafiltration, hemodialysis, intra-aortic balloon pumping or ventricular assist device, etc.
Total intravenous loop diuretic dose per days | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
Change in overall urine output as quantified by the area under the curve (AUC) of daily urine output | From baseline to day 8 or to discharge (in patients discharged earlier than day 8) or to the occurrence of death (in patients dying before day 8)
Absolute change in body weight | From baseline to day 30
Composite of all-cause death or worsening heart failure (HF) | At day 8
  All-cause death is defined as the occurrence of death from any cause.
  Worsening HF is defined as worsening signs and/or symptoms of HF that require an intensification of intravenous therapy for HF or mechanical ventilatory, renal or circulatory support. Such treatment can include the introduction or up-titration of intravenous diuretics, intravenous nitrates, intravenous inotropes, intravenous vasoactive agents or any other intravenous therapy for HF, or institution of mechanical support such as mechanical ventilation, ultrafiltration, hemodialysis, intra-aortic balloon pumping or ventricular assist device, etc.
Composite of all-cause death or total number of heart failure (HF) events | At day 30
  All-cause death is defined as the occurrence of death from any cause.
  HF event is defined as a hospitalization, an Emergency Department visit, an urgent care visit or an outpatient visit with all the following criteria met: hospitalization or visit due to a primary diagnosis of HF or worsening of HF; at least one symptom of HF; at least two physical examination findings of HF or at least one physical examination finding plus one positive diagnostic test of HF; intensification of therapy for HF.
Composite of all-cause death or total number of unplanned rehospitalizations for heart failure (HF) | At day 30
  All-cause death is defined as the occurrence of death from any cause.
  Rehospitalization for HF is defined as an unplanned rehospitalization after discharge due to a primary diagnosis of HF or worsening of HF. The four criteria defining a HF event need to be met also for HF rehospitalization.
All-cause death | At day 30
  All-cause death is defined as the occurrence of death from any cause.
Cardiovascular death | At day 30
  Cardiovascular death is defined as death due to any of the following conditions (as primary cause): HF; myocardial infarction; arrhythmia and conduction system disturbances; cardiac tamponade; cardiovascular hemorrhage, including major or life-threatening bleeding; thromboembolic events; stroke; cardiovascular procedures; acute aortic syndromes; cardiovascular infection and sepsis (e.g., mediastinitis or endocarditis); any other clearly identified cardiovascular cause; sudden, unexpected death; and death of unknown cause.
Total number of heart failure (HF) events | At day 30
  HF event is defined as a hospitalization, an Emergency Department visit, an urgent care visit or an outpatient visit with all the following criteria met: hospitalization or visit due to a primary diagnosis of HF or worsening of HF; at least one symptom of HF; at least two physical examination findings of HF or at least one physical examination finding plus one positive diagnostic test of HF; intensification of therapy for HF.
Total number of unplanned rehospitalizations for heart failure (HF) | At day 30
  Rehospitalization for HF is defined as an unplanned rehospitalization after discharge due to a primary diagnosis of HF or worsening of HF. The four criteria defining a HF event need to be met also for HF rehospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No